CLINICAL TRIAL: NCT06994494
Title: Noninvasive Continuous BP Monitoring in Newborns Based on Pulsatile Signal Morphological Features Using NIRS
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Emily M. Herzberg, MD, Neonatology Attending, Assistant Professor of Pediatrics, Massachusetts General Hospital
Other Study IDs: 2024P000562; 1R21HD117308-01 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Unstable Blood Pressure; Hypotension
Keywords: Non-invasive blood pressure monitoring; Arterial Line; NIRS; wearable device; Cerebral oximetry
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arterial Line Cohort: We will recruit and measure neonates who are between ≥ 24 weeks and < 44 weeks postmenstrual age, undergoing A-line BP monitoring for clinical reasons.
- Cuff Cohort: We will recruit and measure neonates in the same age range as in the A-line cohort who are at risk for unstable blood pressure but without A-line BP monitoring, as long as they can tolerate manual cuff-based BP measurements at intervals of at least 1-4 hours.

SUMMARY:
The goal of this study is to evaluate if a novel near-infrared spectroscopy (NIRS) device can accurately estimate blood pressure in newborns at risk for unstable blood pressure. The main questions it aims to answer are:

* Can NIRS accurately estimate blood pressure when compared to the gold standard, arterial line blood pressure
* Can NIRS accurately estimate blood pressure when compared to infants with cuff blood pressure monitoring

Researchers will compare NIRS-based estimates to arterial line blood pressure readings and manual cuff measurements to optimize and validate the FlexNIRS device for neonates to accurately estimate blood pressure continuously and noninvasively.

Participants will wear a small, noninvasive NIRS sensor on the forehead.

DETAILED DESCRIPTION:
Continuous blood pressure monitoring is important for critically ill newborns to prevent brain injury caused by dysregulated changes in cerebral perfusion. In addition, continuous blood pressure monitoring is beneficial to management of many other conditions in neonates: including hypoxic-ischemic encephalopathy; for monitoring respiratory issues such as respiratory distress syndrome and pulmonary hypertension related to meconium aspiration syndrome; for managing the vascular resistance in conditions like patent ductus arteriosus and congenital heart failures; for ensuring adequate tissue perfusion during critical illness like sepsis and necrotizing enterocolitis (NEC); and for maintaining vascular tone when using inotropes or vasopressors.

The gold standard for continuous BP monitoring in newborns is via arterial line (A-line BP). However, it involves catheterization of the umbilical or a peripheral artery and can lead to complications such as vasospasm, nerve damage, ischemia, thrombosis, and, in severe cases, limb amputation. Due to these risks, A-line BP monitoring is only used when deemed necessary in critically ill neonates.

Existing noninvasive alternatives, including volume-clamp photoplethysmography cuffs, pulse-transit-time, and tonography, are problematic due to large error and safety concerns. They have been validated primarily for adults and are not tailored for neonates who pose unique challenges due to their fragile limbs, underdeveloped vasculature, immature cardiac function, and mean arterial BP often being less than a third of an adult's (30 mmHg).

To address this critical need for accurate, continuous, and noninvasive BP monitoring in newborns, the study team proposes employing a near-infrared spectroscopy (NIRS) technique on the head, focusing on pulsation tones and shapes in cerebral hemodynamics, which are sensitive to BP changes. The team has developed a wearable, battery-operated NIRS device, called FlexNIRS, capable of providing continuous photoplethysmogram (PPG) with a high temporal resolution of 266 Hz. In adults, the team has shown that the time derivative of its optical pulse waveforms d/dt(PPG) is related to pulsatile blood flow, and found strong correlations between specific features of d/dt(NIRS-PPG) and blood pressure changes. Based on these findings, it is hypothesized that NIRS-PPG collected in the brain is most ideal for neonates, especially given their fragile peripheries, and the head site allowing more robust measure of deep brain with less external factors, such as pressure from the sensor itself, room temperature, and extra arterial resistance that builds up in local peripheries. Importantly, the study team has tested the FlexNIRS in a preterm newborn and found pulsatile morphology patterns comparable to those in adults.

The current study aims to validate this novel technique for BP assessment in the newborn population from up to 80 newborns, divided evenly across Massachusetts General Hospital (MGH) and Brigham and Women's Hospital (BWH). Each measurement will involve monitoring infants with one or two FlexNIRS devices for 3-24 hours a day, for at least one day. This data will be used to refine the study team's FlexNIRS-based blood pressure estimation algorithms and correlate results with invasive A-line BP as the gold standard or periodic BP cuff readings performed by clinical staff. This research will provide invaluable data demonstrating method feasibility and initial clinical utility. The successful execution of this aim will guide the study team to a larger clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≥24 & <44 weeks postmenstrual age
* Hospitalization in MGH or BWH newborn service units
* For A-line BP monitoring: Neonates expected to maintain A-line monitoring for at least the next 12 hours
* For non-A-line monitoring: Neonates at risk for unstable blood pressure (e.g. clinical instability or need for inotropes) and no contraindications to manual cuff BP measurements every 1 to 4 hours

Exclusion Criteria:

* Contraindication to FlexNIRS device placement on the scalp/head
* Underlying congenital/genetic anomalies

Ages: 24 Weeks to 44 Weeks | Sex: All
Age Groups: Child
Study Population: The study population will include 80 neonates of ≥24 weeks and <44 weeks postmenstrual age, with or without A-line BP monitoring for clinical reasons. Subjects will be recruited from the Neonatal Intensive Care Unit at MGH and BWH.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
FlexNIRS-based blood pressure estimation | 04/09/2025 - 11/30/2026
  Determine the correlation between FlexNIRS based blood pressure estimation and invasive A-line blood pressure as the gold standard or periodic BP cuff readings performed by clinical staff.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusettes General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Coded and deidentified data may be shared with collaborators outside of Mass General Brigham. All external data sharing will be tracked and logged, and upon request, this information will be readily available to the subjects. The PI will supervise daily lab/team data management and sharing activities, ensuring strict adherence to the data sharing policies outlined by MGB. No identifiable data will be shared or received from collaborators outside of Mass General Brigham.
Supporting Information: CSR
Time Frame: Still finalizing exact timeline.
Access Criteria: Coded and deidentified data may be shared with collaborators outside of Mass General Brigham. No identifiable data will be shared or received from collaborators outside of Mass General Brigham.

REFERENCES:
- [Background] Wu KC, Martin A, Renna M, Robinson M, Ozana N, Carp SA, Franceschini MA. Enhancing diffuse correlation spectroscopy pulsatile cerebral blood flow signal with near-infrared spectroscopy photoplethysmography. Neurophotonics. 2023 Jul;10(3):035008. doi: 10.1117/1.NPh.10.3.035008. Epub 2023 Sep 6. PMID 37680339
- [Background] Wu KC, Tamborini D, Renna M, Peruch A, Huang Y, Martin A, Kaya K, Starkweather Z, Zavriyev AI, Carp SA, Salat DH, Franceschini MA. Open-source FlexNIRS: A low-cost, wireless and wearable cerebral health tracker. Neuroimage. 2022 Aug 1;256:119216. doi: 10.1016/j.neuroimage.2022.119216. Epub 2022 Apr 19. PMID 35452803
- [Background] Boas DA, Strangman G, Culver JP, Hoge RD, Jasdzewski G, Poldrack RA, Rosen BR, Mandeville JB. Can the cerebral metabolic rate of oxygen be estimated with near-infrared spectroscopy? Phys Med Biol. 2003 Aug 7;48(15):2405-18. doi: 10.1088/0031-9155/48/15/311. PMID 12953906
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- [Background] Gonzalez S, Hsieh WT, Chen TP. A benchmark for machine-learning based non-invasive blood pressure estimation using photoplethysmogram. Sci Data. 2023 Mar 21;10(1):149. doi: 10.1038/s41597-023-02020-6. PMID 36944668
- [Background] Troy R, Doron M, Laughon M, Tolleson-Rinehart S, Price W. Comparison of noninvasive and central arterial blood pressure measurements in ELBW infants. J Perinatol. 2009 Nov;29(11):744-9. doi: 10.1038/jp.2009.86. Epub 2009 Jul 16. PMID 19609309
- [Background] Dionne JM. Determinants of Blood Pressure in Neonates and Infants: Predictable Variability. Hypertension. 2021 Mar 3;77(3):781-787. doi: 10.1161/HYPERTENSIONAHA.120.14587. Epub 2021 Feb 10. PMID 33566691
- [Background] Rao A, Eskandar-Afshari F, Weiner Y, Billman E, McMillin A, Sella N, Roxlo T, Liu J, Leong W, Helfenbein E, Walendowski A, Muir A, Joseph A, Verma A, Ramamoorthy C, Honkanen A, Green G, Drake K, Govindan RB, Rhine W, Quan X. Clinical Study of Continuous Non-Invasive Blood Pressure Monitoring in Neonates. Sensors (Basel). 2023 Apr 2;23(7):3690. doi: 10.3390/s23073690. PMID 37050750
- [Background] Alonzo CJ, Nagraj VP, Zschaebitz JV, Lake DE, Moorman JR, Spaeder MC. Blood pressure ranges via non-invasive and invasive monitoring techniques in premature neonates using high resolution physiologic data. J Neonatal Perinatal Med. 2020;13(3):351-358. doi: 10.3233/NPM-190260. PMID 31771082
- [Background] Lynch TM. Invasive and noninvasive pressure monitoring in neonates. J Perinat Neonatal Nurs. 1987 Jul;1(1):58-71. doi: 10.1097/00005237-198707000-00010. No abstract available. PMID 3451967
- [Background] Hahn GH, Hyttel-Sorensen S, Petersen SM, Pryds O, Greisen G. Cerebral effects of commonly used vasopressor-inotropes: a study in newborn piglets. PLoS One. 2013 May 20;8(5):e63069. doi: 10.1371/journal.pone.0063069. Print 2013. PMID 23700412
- [Background] Turner MA, Baines P. Which inotrope and when in neonatal and paediatric intensive care? Arch Dis Child Educ Pract Ed. 2011 Dec;96(6):216-22. doi: 10.1136/adc.2008.143925. Epub 2011 Aug 3. No abstract available. PMID 21813560
- [Background] Rhee CJ, da Costa CS, Austin T, Brady KM, Czosnyka M, Lee JK. Neonatal cerebrovascular autoregulation. Pediatr Res. 2018 Nov;84(5):602-610. doi: 10.1038/s41390-018-0141-6. Epub 2018 Sep 8. PMID 30196311
- [Background] Selb J, Wu KC, Sutin J, Lin PI, Farzam P, Bechek S, Shenoy A, Patel AB, Boas DA, Franceschini MA, Rosenthal ES. Prolonged monitoring of cerebral blood flow and autoregulation with diffuse correlation spectroscopy in neurocritical care patients. Neurophotonics. 2018 Oct;5(4):045005. doi: 10.1117/1.NPh.5.4.045005. Epub 2018 Nov 13. PMID 30450363
- [Background] Sunwoo J, Zavriyev AI, Kaya K, Martin A, Munster C, Steele T, Cuddyer D, Sheldon Y, Orihuela-Espina F, Herzberg EM, Inder T, Franceschini MA, El-Dib M. Diffuse correlation spectroscopy blood flow monitoring for intraventricular hemorrhage vulnerability in extremely low gestational age newborns. Sci Rep. 2022 Jul 27;12(1):12798. doi: 10.1038/s41598-022-16499-3. PMID 35896691